CLINICAL TRIAL: NCT02518256
Title: Lavage of the Uterine Cavity for the Diagnosis of Ovarian and Tubal Carcinoma - Study of Sensitivity and Specificity
Acronym: LUDOC II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Paul Speiser, Prof.MD,, Prof. Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EK 1151/2014
Record Dates: First submitted 2015-06-30; First posted 2015-08-07 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Epithelial Cancer
Keywords: Neoplasms; Glandular and Epithelial; Ovarian Neoplasms; Ovarian cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- (Suspected) Ovarian Epithelial Cancer (Other): Lavage of the Cavum uteri and proximal fallopian tubes
  Interventions: Procedure: Lavage of the Cavum uteri and proximal fallopian tubes

INTERVENTIONS:
Procedure: Lavage of the Cavum uteri and proximal fallopian tubes

SUMMARY:
The ovarian surface, the Fallopian tubes, the uterine cavity and the peritoneal cavity all together form a communicating compartment. The physiologic function of the ciliated lining of the tubes is to transport the egg, after ovulation, into the uterine cavity. Thus, making it very likely that exfoliated cells from pathologic changes of the ovarian surface and Fallopian tube lining will be present in a lavage from the uterine cavity.

The proof of concept that malignant cells from the upper genital tract get transported even into the lower genital tract was recently published by Kind I. et al. Liquid-based cervical cytology allows not only cytological evaluation but also collection of DNA. A panel of genes that are commonly mutated in endometrial and ovarian cancers was assembled with new whole-exome sequencing data from 22 endometrial cancers and previously published data on other tumour types, including mutations in the TP53 gene. This panel was used to search for mutations in 24 endometrial and 22 ovarian cancers and identified mutations in all 46 samples. With a sensitive massively parallel sequencing method, it was possible to identify the same mutations in the DNA from liquid Pap smear specimens in 100% of endometrial cancers (24 of 24) and in 41% of ovarian cancers (9 of 22).

In the current project the investigators will study the specificity and sensitivity of the lavage of uterine cavity and proximal tubes as a test to differentiate between malign and benign ovarian tumours. The investigators aim to detect cells from EOCs or genetic material from those cells in the lavage.

DETAILED DESCRIPTION:
Epithelial ovarian cancer (EOC) is the leading cause of death among gynaecologic malignancies in western civilized countries, with an estimated prevalence in Europe and the US of 752,600 in 2007 and 59,828 deaths annually. Treatment and survival of the patients depend primarily on the stage of the disease. Of all EOC patients only 25% are diagnosed at an early stage while the tumour is confined to the pelvis. In these cases the five-year survival rate is 80% to 90% and the disease can often be cured by the combination of surgery and chemotherapy. Unfortunately, almost 75% of women affected have advanced stage disease with metastatic spread throughout the abdominal cavity or to retroperitoneal lymph nodes at the time of diagnosis; five-year survival rates drop to 10%-30% for advanced disease, despite maximum surgical effort and combination chemotherapy.

Currently, state of the art differential diagnosis between malignant and benign ovarian pathologies suspicious for EOC relies predominantly on transvaginal ultrasonography and serum cancer antigen (CA-125) measurements. The specificity of these diagnostic tools however is low, and both tests are not effective enough to reliably differentiate between benign and malignant conditions. Even in highly specialised units, of all patients receiving surgery for suspected ovarian cancer only about 20% will have a malignant disease. These findings underline the need for new diagnostic tests, able to better differentiate between benign and malignant ovarian changes. This would possibly spear many patients from unnecessary surgery completely and improve the triage of patients with malignant ovarian tumours to highly specialised gynaecologic oncology units.

A promising approach for improvement of differential diagnosis of suspicious ovarian changes has been established by Paul Speiser and Robert Zeillinger (Molecular Oncology Group, Department of General Gynaecology and Gynaecologic Oncology, Medical University of Vienna, Austria) (EK 1148/2011). This approach is called the ALPINE technique (Austrian Lavage Procedure for the Detection of tubal Intraepithelial Neoplasms) (manuscript under preparation). It includes a lavage of the uterine cavity and proximal fallopian tubes and subsequent analysis of this lavage fluid for the presence of pre-malignant and malignant cells.

For the proof of principle that tumour cells are shed from ovarian cancer and can be found in the lavages of the uterine cavity, uterine lavages were collected before a surgical intervention for suspected ovarian malignancy at the investigators' institution and at the Catholic University Leuven, Department of Obstetrics and Gynaecology. After malignancy was confirmed, genetic changes in the TP53 and KRAS gene were determined in tumour tissue. In a set of 9 epithelial ovarian cancer patients (EOC) and 1 ovarian metastases of a signet ring carcinoma, the presence of these genetic changes was examined in lavage samples, using digital droplet PCR (ddPCR). Ten genetic changes were identified in tumour tissue of these patients and 9/10 (90%) of these changes were detected in the corresponding lavage specimen too. Mutation rates were in the range between 0.01% and 39.65% in EOC patients. Furthermore, a filter approach, followed by p53 immunofluorescence staining was established, confirming the presence of tumour cells in the lavage sample of one additional patient.

In a next step, lavage samples of 22 ovarian carcinoma patients, and if applicable corresponding tumour tissue, were analysed through deep sequencing by the group of Bert Vogelstein (Johns Hopkins University, Baltimore, USA). The presence of genetic changes, indicative for ovarian cancer, could be confirmed in 16/22 (72.7%) lavage specimen. Of 18 patients, corresponding tumor tissues were available, showing the same mutation.

These results are proof that ovarian cancer cells are shed into the fallopian tubes and uterine cavity, and can be collected through our ALPINE technique. The fact that ovarian cancer cells were detected with high sensitivity in the lavage of the uterine cavity and proximal tubes shows that this approach has a great potential in differential diagnosis of ovarian masses.

ELIGIBILITY:
Inclusion Criteria:

* suspected ovarian cancer
* verified ovarian cancer

Exclusion Criteria:

* pregnant
* incapacitated persons

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of somatic mutation analysis in at least one of the analyzed genes in cells found in the lavage of the uterine cavity and proximal tubes. | Day 1
  In the current project the investigators will study the specificity and sensitivity of the lavage of uterine cavity and proximal tubes as a test to differentiate between malign and benign ovarian tumours. The investigators aim to detect cells from EOCs by somatic mutation analysis of the genetic material from those cells in the lavage.
  To detect cells from EOCs, analysis of lavage fluid will be carried out applying the sensitive massively parallel sequencing method published by Kinde et al. Mutations in the following genes will be analysed: AKT1, APC, ARID1A, BRAF, CTNNB1, CSMD3, CDKN2A, EGFR, FBXW7, FAT3, FGFR2, KRAS, MLL2, NRAS, PTEN, PIK3CA, PIK3R1, PPP2R1A, PIK3R, RNF43, and TP53.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Speiser, Prof.,Dr.,MD, Principal Investigator — Paul SpeiserMedical University Vienna, Dptm. of Obstetrics & Gynaecology
Locations (4):
- Medical University Vienna, Dptm. of Obstetrics & Gynaecology, Vienna, Austria
- Catholic University Leuven, Leuven, Belgium
- Charles University Pilsen, Pilsen, Czechia
- Klinikum Essen Mitte, Essen, Germany